CLINICAL TRIAL: NCT00710957
Title: Role of Vitamin D Status on Physical Function and Falls in Adults of Advanced Age
Brief Title: Vitamin D and Physical Function in Older Adults
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00005739
Record Dates: First submitted 2008-07-02; First posted 2008-07-08 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Vitamin D; Physical Function
Keywords: Vitamin D; Physical Function; Falls; Aging; CHS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CHS All Stars: CHS All Stars is an ancillary study of the Cardiovascular Health Study (CHS), a longitudinal, observational, population-based study of the onset, progression, and course of heart disease and stroke in the elderly which began in 1988. The All Stars study reexamined the survivors of CHS to determine the likelihood of maintaining function later in life. A focus was to determine whether age-related biological factors are long-term predicators of functional aging which was assessed through a follow-up exam (Yr 18 visit conducted in 2005-06, n=1674 older adults, mean age =84 years) and 3 yrs of subsequent 6 month interval phone contacts. Vitamin D status (serum 25(OH)D and PTH) is being assessed in all CHS All Stars participants who provided a blood sample at the Yr 18 visit (n~1100).

SUMMARY:
Projections from NHANES III indicate that approximately 12,000,000 U.S. adults ≥ 60 years of age have vitamin D insufficiency (serum 25(OH)D < 50 nmol/L). A growing body of evidence suggests that vitamin D status may be important in biologic processes involved in the maintenance of physical function. To test the hypothesis that vitamin D insufficiency is associated with poorer muscle strength and physical performance, we propose to evaluate the role of vitamin D status (serum 25(OH)D) on physical function and falls in the CHS All Stars cohort, a population of advanced age. The specific aims are as follows:

Specific Aim 1. To describe the prevalence and correlates of vitamin D insufficiency in adults of advanced age.

Specific Aim 2. To examine the cross-sectional association between vitamin D status and muscle strength (leg and grip strength), physical performance (3 m/15 ft walk time, repeated chair stands, and standing balance), self-reported physical function (mobility, ADL and IADL disability), and falls.

Specific Aim 3. To examine the longitudinal association between vitamin D status at baseline and incident disability (mobility, ADL and IADL disability) over 3 years of follow-up.

Research Hypotheses: Low vitamin D status (25(OH)D < 50 nmol/L) will be associated with (a) lower levels of muscle strength and physical performance; (b) higher levels of self-reported limitations in physical function and falls; and (c) greater odds of incident disability.

ELIGIBILITY:
Inclusion Criteria:

* Participant in the main CHS study

Exclusion Criteria:

* Not willing to give consent

Min Age: 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Cardiovascular Health Study (CHS), is a longitudinal, observational, population-based study of the onset, progression, and course of heart disease and stroke in the elderly which began in 1988. We are only examining those that participated in the the CHS All Stars which is from the same cohort of people who were still alive in 2005 when enrollment began. We approached everyone who was in the CHS study and asked them to participate in the CHS All Stars study. Blood samples were collected at the year 18 visit and analyzed for serum 25(OH)D.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2008-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To examine the association between vitamin D status and muscle strength (leg, grip strength), physical performance (3m/15 ft walk time, repeated chair stands, and balance), self-reported physical function (mobility, ADL and IADL disability), and falls. | At the year 18 visit of the CHS study
To examine the longitudinal association between vitamin D status at baseline and incident disability (mobility, ADL and IADL disability) over 3 years of follow-up. | Years 18 - 21 of CHS Study

SECONDARY OUTCOMES:
To describe the prevalence and correlates of vitamin D insufficiency in adults of advanced age. | Year 18 of CHS study

CONTACTS AND LOCATIONS:
Overall Officials: Denise Houston, PhD, Principal Investigator — Wake Forest University Health Sciences